CLINICAL TRIAL: NCT04558840
Title: Enhanced Recovery After Bilateral Reduction Mammaplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: interim analysis completed
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey M. Kenkel, Chairman, Department of Plastic Surgery, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STU 2020-0813
Record Dates: First submitted 2020-09-02; First posted 2020-09-22 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Mammaplasty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Enhanced Recovery After Surgery (ERAS) Arm (Active Comparator): ERAS Arm will undergo multimodal regiment:
  Before Surgery- gabepentin 300mg and celecoxib 400mg once the day before surgery and again 3 hours prior to surgery.
  During surgery- subjects will receive ketorolac 30mg IV ketorolac once (15mg for patients age 64 years and above).
  Post-operatively- Gabapentin 100mg three times daily for POD0-7, ketorolac 10mg four times daily for POD1-5 days, and ondansetron 4mg as needed for nausea; patients will also have a prescription for hydrocodone-acetaminophen 5/325mg tabs that they may fill if needed for emergency/breakthrough pain.
  Interventions: Procedure: Macromastia
- Current Practice Arm (Active Comparator): The current practice arm will include: post-operatively, hydrocodone-acetaminophen 5/325mg tabs and ibuprofen 800mg, as needed for pain. Additionally, acetaminophen may be used in conjunction with the above regiment. Ibuprofen and acetaminophen can be taken as needed or alternating every 6 hours, scheduled.
  Interventions: Procedure: Macromastia

INTERVENTIONS:
Procedure: Macromastia — Patients with macromastia seeing the principle investigator (PI) (JMK) at his office at the Outpatient Building, which includes the Outpatient Surgery Center (OSC), in the Department of Plastic Surgery clinic at UT-Southwestern for their initial operative consultation for reduction mammaplasty will be offered enrollment in the trial if they are deemed appropriate surgical candidates, based on the PI's clinical judgement and expertise.
  Other Names: Mammaplasty

SUMMARY:
This single-center, clinical trial is being conducted to determine whether non-narcotic pain regiments are as effective as narcotic-based regiments in reducing post-operative pain in patients undergoing breast reduction in the outpatient setting.

DETAILED DESCRIPTION:
This is a non-blinded, non-inferiority, randomized control trial with the primary outcome of interest being overall pain, with secondary outcomes including adverse effects from pain medications, patient satisfaction with their pain regiment and with their surgery, and the impact of pain on their daily activities. This study is designed to follow one-hundred (100) qualified and consenting patients seeing the PI/surgeon (JMK) at his office at UT Southwestern for their initial operative consultation for macromastia. If patients meet eligibility criteria, they will be offered enrollment in the trial.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing bilateral breast reduction (reduction mammaplasty) with the PI in the outpatient setting
* Age 18 and older
* BMI less than 40, non-smokers.

Exclusion Criteria:

* age less than 18,
* BMI over 40,
* smokers,
* uncontrolled diabetes,
* American Society of Anesthesiologists (ASA) status scores 3 or higher
* patients with allergies to any of the medications in the ERAS or current practice regiments (gabapentin, celecoxib, ketorolac, ondansetron, or hydrocodone).
* History of narcotic or IV drug abuse
* History of chronic pain
* Hypersensitivity or allergy to any of these drugs: gabapentin, celecoxib, ketorolac, hydrocodone, ibuprofen or acetaminophen
* Current pregnancy or planning pregnancy in the next xx weeks/ months
* Contraindications to NSAID drugs (ketorolac, ibuprofen, celecoxib): coagulation disorder, active bleeding, severe renal impairment, hepatic impairment.
* Contraindications to gabapentin: caution for CrCl <60, caution in elderly, caution if alcohol consumption
* Contraindications to acetaminophen: hepatic or renal impairment, chronic alcohol use

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Post-operative Pain Questionnaire | Day 0 - Day 7
  Determine the efficacy of non-narcotic pain regiments in patients undergoing breast reduction surgery and compare it to narcotic-based pain regiments in improving post-operative pain in patients undergoing breast reduction surgery.
  Patients will be asked to rate their pain from a scale of 0 ("No Pain") to 10 ("Pain as bad as you can imagine").

SECONDARY OUTCOMES:
Post operative Patient Satisfaction Questionnaire: Postoperative Reduction Module Satisfaction with Outcome | Day 0- Day 7
  The following questionnaires will be used to track the patients satisfaction following their procedure: BREAST-Q Postoperative Reduction Module Satisfaction with Outcome.
  Patients will be asked to rate their satisfaction with: Very dissatisfied, Somewhat dissatisfied, Somewhat satisfied or very satisfied.
Post operative Patient Satisfaction Questionnaire: Postoperative Module Satisfaction with Information Survey | Day 0- Day 7
  The following questionnaires will be used to track the patients satisfaction following their procedure: BREAST- Q Postoperative Reconstruction Module Satisfaction with Information Survey.
  Patients will be asked to rate their satisfaction with: Very dissatisfied, Somewhat dissatisfied, Somewhat satisfied or very satisfied.
Post operative Quality of Life Questionnaire | Day 0- Day 7
  The following questionnaires will be used to track the patients satisfaction following their procedure.
  The postoperative questions do not have an applicable scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Kenkel, Principal Investigator — UT Southwestern
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States